CLINICAL TRIAL: NCT05808231
Title: An aDaptive, multicEnter, rAndomized, Open-Label, Controlled Trial to Assess Effectiveness and Safety of Quinine Sulfate for COVID-19 in Hospitalized Adults
Brief Title: Effectiveness and Safety of Quinine Sulfate as add-on Therapy for COVID-19 in Hospitalized Adults in Indonesia ( DEAL-COVID19 )
Acronym: DEAL-COVID19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Padjadjaran (Other)
Collaborators: National Research and Innovation Agency of Indonesia (Unknown); Prodia Diacro Laboratories P.T. (Industry)
Responsible Party: Principal Investigator, Keri Lestari, Prof. Dr. Keri Lestari, M.Si, S.Si, Apt., Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pharm-202005.12
Record Dates: First submitted 2023-04-10; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19; Quinine Sulfate
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Quinine

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to be in Arm 1 or Arm 2 using pre-defined randomisation list; 1:1 for each arm.
  Arm 1 receives Standard of Care Arm 2 receives Standard of Care+Quinine Sulfate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Standard of Care alone
  Interventions: Drug: Standard of Care
- Experimental Group (Other): Standard of Care + Quinine Sulfate
  Interventions: Drug: Standard of Care + Quinine Sulfate

INTERVENTIONS:
Drug: Standard of Care + Quinine Sulfate — Standard of Care + Quinine Sulfate
  Arms: Experimental Group
Drug: Standard of Care — Standard of Care for COVID-19 mild and moderate symptom
  Arms: Control Group

SUMMARY:
This is a multicenter, randomized, open-label, controlled trial to evaluate the effectiveness and safety of Quinine Sulfate as an add-on therapy in hospitalized adults with COVID-19.

The study is a multi-center trial that will be conducted in up to approximately 2 sites nationally. New sites may be added as needed after appropriate assessment. Interim monitoring will be conducted to evaluate the arms and for safety and effectiveness. Any changes would be accompanied by an updated sample size.

Subjects will be assessed while hospitalized. All subjects will undergo a series of laboratory tests (CBC, SGOT, SGPT, Ureum, Creatinine, EKG, and PCR), clinical examination (clinical assessment, vital signs, accompanying drugs, and other medical conditions) and safety assessment (serious adverse events/ SAE)

Randomization will be performed 1:1 for each arm. Arm 1 = Standard of Care (SoC) alone, arm 2 = SoC + Quinine Sulfate

DETAILED DESCRIPTION:
This is an adaptive, multicenter, randomized, open-label, controlled trial to evaluate the effectiveness and safety of quinine sulfate in mild to moderate COVID-19 hospitalized adults with confirmed positive Rapid Test or PCR.

The study is a multi-center trial that will be conducted in up to approximately 2 sites nationally. New sites may be added as needed after appropriate assessment. Interim monitoring will be conducted to evaluate the arms and for effectiveness and safety. Any change would be accompanied by an updated sample size.

Eligible patients are male and female patients aged ≥ 18 years to < 60 years old who are hospitalized with Covid-19 based on clinical symptoms determined by physician and confirmed by Rapid Test or PCR test with mild to moderate symptoms that fulfill the inclusion and exclusion criteria stated in the protocol. Total Subjects: 100

Subjects with any of these conditions will be excluded:

* Received quinine sulfate, hydroxychloroquine, chloroquine, lumefantrine, or mefloquine within 30 days prior to this research;
* Having receive any treatment for COVID-19 prior to this research;
* Any contraindication to quinine sulfate
* Inability to swallow pills or any other reason that compliance with the medical regimen is not likely;
* Pregnant and breastfeeding;
* Severe underlying disease where treatment and follow up is not likely to be beneficial to the patient based on physician judgement (e.g. retinopathy, cardiovascular disease (QTc > 500 mdet (narrow QRS); QTc ≥ 550 mdet (wide QRS)), heart arrythmia, uncontrolled diabetes mellitus, hypertension, chronic pulmonary disease, asthma, chronic kidney disease (Creatinine > 2x normal value), liver disease (SGOT/SGPT > 2x normal value), chronic neurological disease, or etc.). This includes people requiring care in designated supported living facilities and severe dementia;
* Platelet count less than 150,000 and more than 450,000 cells/μL;
* Possibility of being transferred to a non-study-hospital within 72 hours.

Any suspected serious adverse event reaction is reported to CRO/Sponsor and EC within 24 hours, using patient's study ID.

During the study conduct, the study team shall keep all the relevant source documents and transcribe the data in case report form (CRF). The study team should also update study essential document (e.g. subject log, investigational product accountability log, etc.) and keep the copy captured by scan/camera for monitoring/audit/inspection purpose.

The study is expected to be finished in 1,5 years.

Standard of Care (SoC) treatment is based on COVID-19 Treatment Protocol (4th edition, 2020) published by Medical Associations (PDPI, PERKI, PAPDI,PERDATIN, IDAI).

MILD CASE:

Arm 1 = SoC alone Arm 2 = SoC + Quinine Sulfate (2 tablets of Quinine Sulfate 200 mg administered orally once daily for 5 days).

MODERATE CASE:

Arm 1 = SoC alone Arm 2 = SoC + Quinine Sulfate (2 tablets of Quinine Sulfate 200 mg administered orally every 12 hours in Day 1, followed with 2 tablets of Quinine Sulfate 200 mg administered once daily for 5-7 days).

It is anticipated that patients with COVID-19 will present to participating hospitals, and that no external recruitment efforts towards potential subjects are needed. Recruitment efforts may also include dissemination of information about this trial to other medical professionals/hospitals.

The Ethics Committee will approve the recruitment process and all materials prior to any recruitment to prospective subjects directly.

Screening will begin with a brief discussion with study staff. Some will be excluded based on demographic data and medical history (i.e., pregnant, < 18 years of age, renal failure, etc.). Information about the study will be presented to potential subjects (or legally authorized representative) and questions will be asked to determine potential eligibility. Screening procedures can begin only after informed consent is obtained.

To evaluate the effectiveness of Quinine Sulfate in the therapy of mild to moderate hospitalized adults with confirmed COVID-19 based on subject's clinical condition assessed using a 7-point ordinal scale. Secondary parameters will be Incidence and duration of Oxygenation (days of oxygenation), incidence is defined as number of days from randomization until the subject received oxygenation, duration is defined as total days of the use of oxygenation; incidence of Ventilation (days to receiving ventilation) and length of stay in hospital (after subject received randomization code until subject discharge/death/recovered).

To evaluate the safety of quinine sulfate on laboratory parameters, serious adverse events and QT interval based on ECG result.

* Change in CBC, SGOT, SGPT, Ureum and Creatinine;
* Number of reported Serious Adverse Event (SAE);
* Change in QT interval based on ECG result.

Analyses relate outcome to the randomly allocated treatment (e.g. intent-to-treat). The primary analyses assess any effects of treatment allocation on all-cause in-hospital mortality, analyzing separately people who already at mild and moderate level at entry and those who did not. Interim analysis will be carried out after 50% subject enrolled. A Data Safety Monitoring Board (DSMB) will monitor ongoing results to ensure subject well-being and safety as well as study integrity. The DSMB will evaluate the study safety parameter after 50% subject enrolled in the study.

The main secondary analyses assess any effects of treatment allocation on:

* Duration of hospitalization (time from randomization to discharge) (days);
* Incidence and duration of Oxygenation;
* Incidence and duration of Ventilation;
* Clinical outcome from baseline at day 10 or if discharged earlier

Study related data will be recorded in electronically. All the data in the source documents shall be collected by the study team to be transcribed in the electronic case report form (eCRF) and other study documents are stored in the electronic trial master file (eTMF). Once the document recorded, the electronic data will be automatically available for monitoring/audit/inspection purpose. All the electronic system used and data recording in the study must be conducted in compliance to Good Clinical Practice.

The investigator must assure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On CRFs or other documents submitted to the funder, subjects should not be identified by their names, but by an identification code. The investigator should keep a subject enrolment log showing codes, names and addresses. The investigator should maintain documents not for submission to funder, e.g. subjects' written consent forms, in strict confidence.

The investigator shall ensure the quality control and quality assurance of the data generated during the study and how the data will be handled, including providing access to monitoring activities, audit and inspection and source documents which will be used in the study. Investigator will permit monitoring, audits and inspections by funder/CRO, EC, and regulatory bodies.

All source records including electronic data (if any) will be stored in secured systems in accordance with institutional policies and locally applicable regulation. All the essential documents should be retained until at least 5 years after the study ended or based on the applicable regulatory requirements or based on the agreement with the funder.

The Drug Safety Monitoring Board (DSMB) is an Independent Data Monitoring Committee consisting of doctors who are experienced in clinical trials, statisticians, and other members who do not direct involvement with this study. The DSMB responsible for the ongoing review of a clinical trial and for making recommendations to the sponsor concerning the continuation, modification, and termination of the trial as it is being conducted. The DSMB will be the only committee that is allowed to review the confidential data in the study. The statistician will analyze the subject's security data and report to DSMB to be evaluated more closely. The key responsibilities of the DSMB are to ensure patient safety by routine review of overall safety data including all SAEs, SUSARs, all severe AEs and AEs leading to drug or study discontinuation and, where applicable, literature cases and information from Competent Authorities(CAs) and by judging the relevance of the events for patients' safety. The DSMB will review the results of data that has been analyzed in accordance with SAP and consider other evidence arising from other studies and will provide advice to the Trial Steering Committee (TSC) (the research committee and national coordinator) regarding the sustainability of this study. The DSMB may recommend the TSC to the recruitment or study termination or provide recommendations related to alternatives treatment (if any)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥ 18 years to 50 years old who are hospitalized with Covid-19 based on clinical symptoms determined by physician and confirmed by Rapid Test or PCR test with mild to moderate symptoms
* Female subjects of child-bearing age agree to take effective contraceptive measures during the study until seven days of the last oral medication
* Willing to receive a random assignment to any designated treatment group and not participating in another study at the same time
* Not participating in other research at the same time.
* Subjects agreed to participate in the study and signed an information sheet and informed consent.

Exclusion Criteria:

* Received quinine sulfate, hydroxychloroquine, chloroquine, lumefantrine, or mefloquine within 30 days prior to this research;
* Having receive any treatment for COVID-19 prior to this research;
* Any contraindication to quinine sulfate
* Inability to swallow pills or any other reason that compliance with the medical regimen is not likely;
* Pregnant and breastfeeding;
* Severe underlying disease where treatment and follow up is not likely to be beneficial to the patient based on physician judgement (e.g. retinopathy, cardiovascular disease (QTc > 500 mdet (narrow QRS); QTc ≥ 550 mdet (wide QRS)), heart arrythmia, uncontrolled diabetes mellitus, hypertension, chronic pulmonary disease, asthma, chronic kidney disease (Creatinine > 2x normal value), liver disease (SGOT/SGPT > 2x normal value), chronic neurological disease, or etc.). This includes people requiring care in designated supported living facilities and severe dementia;
* Platelet count less than 150,000 and more than 450,000 cells/μL;
* Possibility of being transferred to a non-study-hospital within 72 hours.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
The clinical condition of the subjects assessed on a 7-point ordinal scale | From the date of randomization until the date of first documented subject discharge or death from any cause, assessed up to 10 days
  The clinical condition of the subjects was assessed until day 10 using a 7-point ordinal scale, as follows:
  1. Death
  2. Hospitalization, with invasive mechanical ventilation or ECMO
  3. Hospitalization, with non-invasive ventilation or high-flow oxygen device;
  4. Hospitalized, requires additional oxygen;
  5. Hospitalized, does not require additional oxygen;
  6. Not hospitalized, activity restrictions;
  7. No hospitalization, no activity restrictions

SECONDARY OUTCOMES:
Duration of oxygenation | From the date of randomization until the date of first documented subject discharge or death from anycause, assessed up to 10 days
  Total days of oxygen supplementation
Duration of ventilation | From the date of randomization until the date of first documented subject discharge or death from anycause, assessed up to 10 days
  Total days of receiving ventilation
Length of stay | From the date of randomization until the date of first documented subject discharge or death from anycause, assessed up to 10 days
  Total days the subjects were hospitalized

OTHER OUTCOMES:
Safety Outcome (Change in CBC, SGOT, SGPT, Ureum and Creatinine) | Will be examined at days 0 (before treatment) and at the end of treatment
  Change in CBC, SGOT, SGPT, Ureum and Creatinine on the day before treatment and at the end of treatment/on discharge from the hospital
Safety Outcome (Number of reported Serious Adverse Event) | From the date of randomization until the date of first documented subject discharge or death from anycause, assessed up to 10 days
  Number of reported Serious Adverse Event
Safety Outcome (Change in QT interval based on ECG result) | Will be examined at days 0, 3, 6, 9 after starting treatment
  Change in QT interval based on ECG results measured on days 0, 3, 6 and 9 after starting treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Gatot Soebroto Army Central Hospital (RSPAD), Jakarta, DKI Jakarta
  - Dr. Hasan Sadikin Central General Hospital (RSHS), Bandung, West Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mehra MR, Desai SS, Ruschitzka F, Patel AN. RETRACTED: Hydroxychloroquine or chloroquine with or without a macrolide for treatment of COVID-19: a multinational registry analysis. Lancet. 2020 May 22:S0140-6736(20)31180-6. doi: 10.1016/S0140-6736(20)31180-6. Online ahead of print. PMID 32450107
- [Result] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Result] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Result] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Result] Colson P, Rolain JM, Raoult D. Chloroquine for the 2019 novel coronavirus SARS-CoV-2. Int J Antimicrob Agents. 2020 Mar;55(3):105923. doi: 10.1016/j.ijantimicag.2020.105923. Epub 2020 Feb 15. No abstract available. PMID 32070753
- [Result] Lu H. Drug treatment options for the 2019-new coronavirus (2019-nCoV). Biosci Trends. 2020 Mar 16;14(1):69-71. doi: 10.5582/bst.2020.01020. Epub 2020 Jan 28. PMID 31996494
- [Result] Zhou N, Pan T, Zhang J, Li Q, Zhang X, Bai C, Huang F, Peng T, Zhang J, Liu C, Tao L, Zhang H. Glycopeptide Antibiotics Potently Inhibit Cathepsin L in the Late Endosome/Lysosome and Block the Entry of Ebola Virus, Middle East Respiratory Syndrome Coronavirus (MERS-CoV), and Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV). J Biol Chem. 2016 Apr 22;291(17):9218-32. doi: 10.1074/jbc.M116.716100. Epub 2016 Mar 7. PMID 26953343
- [Result] Rainsford KD, Parke AL, Clifford-Rashotte M, Kean WF. Therapy and pharmacological properties of hydroxychloroquine and chloroquine in treatment of systemic lupus erythematosus, rheumatoid arthritis and related diseases. Inflammopharmacology. 2015 Oct;23(5):231-69. doi: 10.1007/s10787-015-0239-y. Epub 2015 Aug 6. PMID 26246395
- [Result] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Result] Zhou D, Dai SM, Tong Q. COVID-19: a recommendation to examine the effect of hydroxychloroquine in preventing infection and progression. J Antimicrob Chemother. 2020 Jul 1;75(7):1667-1670. doi: 10.1093/jac/dkaa114. PMID 32196083
- [Result] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Result] Chen J, Liu D, Liu L, Liu P, Xu Q, Xia L, Ling Y, Huang D, Song S, Zhang D, Qian Z, Li T, Shen Y, Lu H. [A pilot study of hydroxychloroquine in treatment of patients with moderate COVID-19]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2020 May 25;49(2):215-219. doi: 10.3785/j.issn.1008-9292.2020.03.03. Chinese. PMID 32391667
- [Result] Lestari K, Sitorus T, Instiaty, et al. (last). Molecular docking of quinine, chloroquine and hydroxychroloquine to angiotensin converting enzyme 2 (ACE2) for discovering new potential COVID-19 antidote. J Adv Pharm Edu Res. 2020;10(2):1-4.
- [Result] Mauthe M, Orhon I, Rocchi C, Zhou X, Luhr M, Hijlkema KJ, Coppes RP, Engedal N, Mari M, Reggiori F. Chloroquine inhibits autophagic flux by decreasing autophagosome-lysosome fusion. Autophagy. 2018;14(8):1435-1455. doi: 10.1080/15548627.2018.1474314. Epub 2018 Jul 20. PMID 29940786
- [Result] Biot C, Daher W, Chavain N, Fandeur T, Khalife J, Dive D, De Clercq E. Design and synthesis of hydroxyferroquine derivatives with antimalarial and antiviral activities. J Med Chem. 2006 May 4;49(9):2845-9. doi: 10.1021/jm0601856. PMID 16640347
- [Result] Bray PG, Mungthin M, Hastings IM, Biagini GA, Saidu DK, Lakshmanan V, Johnson DJ, Hughes RH, Stocks PA, O'Neill PM, Fidock DA, Warhurst DC, Ward SA. PfCRT and the trans-vacuolar proton electrochemical gradient: regulating the access of chloroquine to ferriprotoporphyrin IX. Mol Microbiol. 2006 Oct;62(1):238-51. doi: 10.1111/j.1365-2958.2006.05368.x. Epub 2006 Aug 31. PMID 16956382
- [Result] Nqoro X, Tobeka N, Aderibigbe BA. Quinoline-Based Hybrid Compounds with Antimalarial Activity. Molecules. 2017 Dec 19;22(12):2268. doi: 10.3390/molecules22122268. PMID 29257067
- [Result] Graves PR, Kwiek JJ, Fadden P, Ray R, Hardeman K, Coley AM, Foley M, Haystead TA. Discovery of novel targets of quinoline drugs in the human purine binding proteome. Mol Pharmacol. 2002 Dec;62(6):1364-72. doi: 10.1124/mol.62.6.1364. PMID 12435804
- [Result] Kwiek JJ, Haystead TA, Rudolph J. Kinetic mechanism of quinone oxidoreductase 2 and its inhibition by the antimalarial quinolines. Biochemistry. 2004 Apr 20;43(15):4538-47. doi: 10.1021/bi035923w. PMID 15078100
- [Result] Gachelin G, Garner P, Ferroni E, Trohler U, Chalmers I. Evaluating Cinchona bark and quinine for treating and preventing malaria. J R Soc Med. 2017 Feb;110(2):73-82. doi: 10.1177/0141076816688411. No abstract available. PMID 28169590
- [Result] Winstanley, P. Handbook of drugs for tropical parasitic infections. 2nd Edition. Transactions of the Royal Society of Tropical Medicine and Hygiene; 1996.
- [Result] Große M, Ruetalo N, Businger R, Rheber S, Setz C, Auth J, et al. Evidence That Quinine Exhibits Antiviral Activity against SARS-CoV-2 Infection In Vitro. 2020;14.
- [Result] Burhan E, Susanto A, Nasution S, Ginanjar E, Pitoyo C, Susilo A, et al. COVID-19 PROTOCOL. 1st ed. Jakarta: Association of Indonesian Pulmonary Doctors (PDPI); 2020.
- [Result] BPOM. Information on Drugs for COVID-19 in Indonesia
- [Result] WHO. Public health emerging solidarity trial: World Health Organization COVID-19 Core Protocol. 2020.
- [Result] Whitehead J. Sample size calculations for ordered categorical data. Stat Med. 1993 Dec 30;12(24):2257-71. doi: 10.1002/sim.4780122404. PMID 8134732
- See also: Infeksi Emerging: Media Informasi Resmi Terkini Penyakit Infeksi Emerging. — https://infeksiemerging.kemkes.go.id/
- See also: Letter of Recommendation for the Use of Hydroxychloroquine/Chloroquine Phosphate in the Treatment of COVID-19 dated 04 June 2020. — https://www.papdi.or.id/pdfs/886/SURAT%20Rekomendasi%205op%20HCQ_CQ%20(1).pdf
- See also: National Library of Medicine — https://clinicaltrials.gov/
- See also: FDA Drug Safety Communication: New risk management plan and patient Medication Guide for Qualaquin (quinine sulfate) — https://www.fda.gov/drugs/postmarket-drug-safety-information-patients-and-providers/fda-drug-safety-communication-new-risk-management-plan-and-patient-medication-guide-qualaquin/